CLINICAL TRIAL: NCT03700736
Title: Delivering a Post-Partum Weight Loss Intervention Via Facebook vs In-Person Groups: a Feasibility Trial
Brief Title: The Healthy Moms Study: Comparison of a Post-Partum Weight Loss Intervention Delivered Via Facebook or In-Person Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Massachusetts, Worcester (Other); Worcester Polytechnic Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Molly Waring, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H17-206; R34HL136979 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-10-09 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Weight Loss; Diet Modification; Physical Activity
Keywords: post-partum women; social media; Facebook; digital health
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook (Active Comparator): Women will receive the Healthy Moms intervention, a 6-month behavioral weight loss intervention, via a private ("secret") Facebook group. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based lifestyle intervention. A study counselor will facilitate discussions about the topics posted in the Facebook group. Each participant will get an individualized calorie and physical activity goal to help them achieve a healthy weight loss of 1-2 pounds per week. Participants will be encouraged to increase physical activity to 150 minutes per week of moderate intensity activity. Participants will also be encouraged to download the MyFitnessPal app to track daily diet.
  Interventions: Behavioral: Healthy Moms
- Traditional (Active Comparator): Women will receive the Healthy Moms intervention, a 6-month behavioral weight loss intervention, via in-person 90-minute group sessions (weekly in months 1-4, every other week in months 5-6). The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based lifestyle intervention. Intervention components will be introduced in the format of handouts, group discussions, and lists of existing resources. Each participant will get an individualized calorie and physical activity goal to help them achieve a healthy weight loss of 1-2 pounds per week. Participants will be encouraged to increase physical activity to 150 minutes per week of moderate intensity activity. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet.
  Interventions: Behavioral: Healthy Moms

INTERVENTIONS:
Behavioral: Healthy Moms — The 6-month intervention will include dietary and exercise counseling and tips to help participants meet their healthy lifestyle goals. Participants will receive personalized calorie and physical activity goals to help them achieve a healthy weight loss of 1-2 pounds per week. Participants will be encouraged to increase physical activity to 150 minutes per week of moderate intensity activity. Counselors will encourage and support participants to make a plan for incorporating regular physical activity into their lives in a way (i.e., duration per session, frequency per week) that works for that individual woman. We will encourage participants to track their diet and exercise daily. We will encourage participants to use My Fitness Pal to track their diet and activity.

SUMMARY:
The goal of the project is to conduct a feasibility pilot randomized trial comparing delivery of a post-partum weight loss intervention via Facebook versus via in-person group sessions. The project will provide preliminary data needed to finalize the design of a large randomized trial to compare the non-inferiority and cost-effectiveness of the post-partum weight loss intervention delivered via Facebook versus in-person group sessions. If efficacious and cost-effective, the Facebook-delivered intervention leads naturally to strategies for scaling up for widespread impact.

DETAILED DESCRIPTION:
Post-partum weight retention contributes to obesity for many women, increasing risk for cardiovascular disease and other chronic diseases and complicating future pregnancies. Lifestyle interventions have shown to be modestly efficacious for post-partum weight loss in randomized controlled trials, yet interventions with numerous visits are logistically challenging for many post-partum women. Innovative and efficacious treatment models for post-partum weight loss that fit into the busy lives of new moms are needed, and cost-effectiveness is critical for adoption. Facebook may be an efficient platform for delivering evidence-based weight loss programming to post-partum women. Delivering interventions via Facebook allows us to connect with post-partum women where they are, more fully integrating into their lives and daily routines. Investigators have developed a post-partum weight loss intervention based on the Diabetes Prevention Program, tailored to needs of post-partum women and for delivery via Facebook. Investigators will conduct a feasibility pilot randomized trial comparing delivery of a post-partum weight loss intervention via Facebook to in-person group sessions. Primary outcomes are the feasibility of recruitment, sustained participation, contamination, retention, and feasibility of assessment procedures in both treatment conditions. Weight loss will be described as an exploratory outcome. The project will provide preliminary data needed to finalize the design of a large randomized trial to compare the non-inferiority and cost-effectiveness of the post-partum weight loss intervention delivered via Facebook versus in-person group sessions. Demonstrating cost-effectiveness in addition to efficacy of our Facebook-delivered post-partum weight loss intervention is critical to support widespread implementation.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years or older
* 8 weeks to 12 months post-partum at enrollment
* overweight or obese (BMI ≥ 25 kg/m2) per measured height and weight at the baseline visit
* owns a scale
* comfortable reading and speaking in English
* owns an iPhone or Android smartphone
* active Facebook user
* medical clearance (e.g., from primary care provider or obstetrician/gynecologist)
* willing and able to participate in either treatment condition (Facebook or in-person)
* available to attend in-person meetings over the 6-month study period
* 45 minutes or less to travel to intervention meetings
* willing and able to provide informed consent

Exclusion Criteria:

* UConn employee or student who is key personnel on the study, UConn employee or student who is a spouse, dependent, or relative of any key personnel, or UConn student who key personnel on this study teaches
* women who are currently pregnant or plan to conceive during study period
* current participation in clinical weight loss program
* Type 1 or Type 2 diabetes
* medical conditions affecting weight
* medications affecting weight
* incapable of walking 1/4 of a mile without stopping
* pain that prevents engagement in exercise
* previous bariatric surgery
* planned surgery during study period
* plans to move out of the area during the study period
* high depressive symptoms or suicidal ideation
* positive screen for binge eating disorder
* failure to complete the baseline survey
* failure to complete the orientation webinar

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly E. Waring, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waring ME, Libby BA, Moore Simas TA, Bracken ML, Bibeau JL, Herrera V, Wang J, Pagoto SL. Delivering a Post-Partum Weight Loss Intervention via Facebook or In-Person Groups: Protocol for a Randomized Feasibility Pilot Trial. JMIR Res Protoc. 2019 Nov 28;8(11):e15530. doi: 10.2196/15530. PMID 31778116
- [Derived] Waring ME, Pagoto SL, Moore Simas TA, Blackman Carr LT, Eamiello ML, Libby BA, Rudin LR, Heersping GE. Delivering a Postpartum Weight Loss Intervention via Facebook or In-Person Groups: Results From a Randomized Pilot Feasibility Trial. JMIR Mhealth Uhealth. 2023 Apr 27;11:e41545. doi: 10.2196/41545. PMID 37103991

RESULTS

PARTICIPANT FLOW:
Groups:
- Facebook: 6-month post-partum weight loss intervention delivered via a private Facebook group
- Traditional: 6-month post-partum weight loss intervention delivered via in-person group meetings
Period: Overall Study
Arm/Group | Facebook | Traditional
Started (Intervention) | 30 | 32
Completed | 27 | 25
Not Completed | 3 | 7
Not completed — Pregnancy | 1 | 1
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Facebook | Traditional | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (3.5) | 32.3 (4.4) | 32.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 26 | 26 | 52
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants] — greater Hartford, CT region
  participants
    United States | 30 | 32 | 62
Weight [Median (Inter-Quartile Range); unit: pounds] — Weight measured at baseline (pounds)
  pounds | 188.9 [171.0 to 225.3] | 180.6 [168.6 to 214.6] | 186.0 [169.2 to 217.1]

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: Recruitment rates will be calculated from the number of patients approached, screened, consented, and randomized.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Individuals Contacted: Individuals who expressed interest in study participation
Arm/Group | Individuals Contacted
Number analyzed (Participants) | 606
Participants
  Could not reach to screen | 163
  Not interested in participating | 105
  Ineligible at initial eligibility screening | 195
  Eligible but did not complete baseline visit | 65
  Eligible at screening but met additional exclusion criteria or did not complete baseline procedures | 16
  Randomized | 62

2. Primary Outcome: Sustained Participation
Description: We will calculate sustained participation as time to last intervention session attended in the in-person condition and as time to last post, comment, or reaction (based on date of last post or comment reacted to) in the Facebook condition.
Time Frame: 6 months
Population: Latest treatment module participated in based on last intervention meeting attended (Traditional) or last treatment module engaged in based on original posts, replies/comments, reactions, and poll votes (Facebook)
Measure: Median (Inter-Quartile Range); unit: latest treatment module participated in
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
latest treatment module participated in | 20 [19 to 20] | 18 [2 to 20]

3. Primary Outcome: Contamination
Description: Participants in both treatment conditions will report if they have participated in other weight loss programs (online or in-person), and whether they have searched for weight loss support on Facebook or other online social networks.
Time Frame: 6 months
Population: Participants reported use of other weight loss programs and seeking weight loss info/support on social media on the 6-month survey. We report the number and percentage of participants in each condition that reported use of other weight loss programs, sought weight loss info/support on social media, both, or neither. These data are available only for participants who completed the 6-month survey. Note that we encouraged participants in both groups to reference online resources (e.g., recipes).
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 26 | 28
Participants
  Used other weight loss programs & sought weight loss info/support on social media | 1 | 1
  Used other weight loss programs | 3 | 0
  Sought weight loss info or support on social media | 8 | 15
  Neither | 14 | 12

4. Primary Outcome: Retention
Description: Retention is calculated as the percentage of participants who complete the 6-month follow-up study assessment in each condition.
Time Frame: 6 months
Population: Retention is defined as completing 6-month follow-up study assessment (providing weight and/or completing the follow-up survey)
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
Participants
  Retained | 27 | 30
  Lost to follow-up | 3 | 2

5. Primary Outcome: Retention
Description: Retention is calculated as the percentage of participants who complete the 12-month follow-up study assessment in each condition.
Time Frame: 12 months
Population: Retention is defined as completing 12-month follow-up study assessment (providing weight and/or completing the follow-up survey)
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
Participants
  Retained | 28 | 30
  Lost to follow-up | 2 | 2

6. Primary Outcome: Degree of Missingness in Study Measures
Description: Percent of participants missing data on each measure/item included in data collection at baseline.
Time Frame: Baseline
Population: Missing (or incomplete) measures needed for cost-effectiveness aim of subsequent efficacy trial: weight and/or quality of life measure.
Measure: Count of Participants; unit: Participants
Groups:
- Facebook: 6-month behavioral weight loss intervention delivered via a private Facebook group
- Traditional: 6-month behavioral weight loss intervention delivered via in-person group meetings
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
Participants
  Missing (or incomplete) quality of life | 4 | 2
  Available information on both weight and quality of life | 26 | 30

7. Primary Outcome: Degree of Missingness in Study Measures
Description: Percent of participants missing data on each measure/item included in data collection at 6 months.
Time Frame: 6 months
Population: Missing (or incomplete) measures needed for cost-effectiveness aim of subsequent efficacy trial: weight and/or quality of life measure. Note that as quality of measure was assessed as part of 6-month survey, participants who did not complete the survey are missing this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
Participants
  Missing weight and quality of life | 3 | 2
  Missing quality of life | 1 | 3
  Available information on both weight and quality of life | 26 | 27

8. Primary Outcome: Degree of Missingness in Study Measures
Description: Percent of participants missing data on each measure/item included in data collection at 12 months.
Time Frame: 12 months
Population: Missing (or incomplete) measures needed for cost-effectiveness aim of subsequent efficacy trial: weight and/or quality of life measure. Note that as quality of measure was assessed as part of 12-month survey, participants who did not complete the survey are missing this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 30 | 32
Participants
  Missing weight and quality of life | 2 | 2
  Missing quality of life | 0 | 1
  Available information for both weight and quality of life | 28 | 29

9. Secondary Outcome: Weight Change (Exploratory)
Description: Weight will be measured at baseline and 6 months. Percent weight change will be calculated.
Time Frame: 6 months
Population: Percent weight change from baseline to 6 months. All baseline weights were measured at a study visit. At 6 months, weight was measured at a study visit or participants self-reported current or pre-pregnancy weight (if pregnant). Note that due to COVID19, all follow-up weights for wave 2 were self-reported. Complete case weight change is reported.
Measure: Mean (Standard Deviation); unit: percent weight loss from baseline
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 27 | 30
percent weight loss from baseline | -3.0 (7.2) | -5.4 (6.8)

10. Secondary Outcome: Weight Change (Exploratory)
Description: Weight will be measured at baseline and 12 months. Percent weight change will be calculated.
Time Frame: 12 months
Population: Percent weight change from baseline to 12 months. All baseline weights were measured at study visit. At 12 months, weight was measured at study visit or participants self-reported current or pre-pregnancy weight (if pregnant). Note that due to COVID19, all follow-up weights for wave 2 were self-reported. Complete case weight change is reported.
Measure: Mean (Standard Deviation); unit: percent weight loss from baseline
Arm/Group | Facebook | Traditional
Number analyzed (Participants) | 28 | 30
percent weight loss from baseline | -2.8 (7.4) | -4.8 (7.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the intervention and at 6-month and 12-month follow-up assessments
Description: Adverse events were spontaneous reported by participants during the intervention and at follow-up assessments. Depressive symptoms and pregnancy were queried at the 6-month and 12-month assessments.
Arm/Group | Facebook | Traditional
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 25/30 | 23/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Facebook (N=30) | Traditional (N=32)
Communicable disease (e.g., cold, flu) (General disorders) | 15 (17) | 15 (17)
5% or greater weight gain (General disorders) | 2 (2) | 3 (3)
Musculoskeletal pain or injury (not related to exercise) (Injury, poisoning and procedural complications) | 5 (5) | 4 (5)
Pregnancy during intervention or follow-up (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Depressive symptoms (Psychiatric disorders) | 12 (13) | 5 (6)

LIMITATIONS AND CAVEATS:
In wave 2, due to safety concerns related to COVID-19, the last two intervention meetings for the Traditional condition were held via WebEx (vs in-person meetings) and 6-month and 12-month assessments for participants in both conditions were held remotely (vs in-person study visits). Thus in wave 2, all follow-up weights are self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03700736/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03700736/SAP_001.pdf
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03700736/ICF_002.pdf